CLINICAL TRIAL: NCT00138112
Title: Randomized Trial of Prophylactic Versus Empirical Vancomycin for the Prevention of Early Viridans Streptococcal Sepsis After Hematopoietic Cell Transplantation
Brief Title: Trial of Prophylactic Versus Empirical Vancomycin for the Prevention of Streptococcal Sepsis After Hematopoietic Cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03-142
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Streptococcal Sepsis; Hematologic Malignancies
Keywords: Streptococcal Sepsis; Hematopoietic Stem Cell Transplantation; Hematologic Malignancies; Streptococci; Transplant
MeSH Terms: conditions — Hematologic Neoplasms

INTERVENTIONS:
Drug: Empirical Vancomycin
Drug: Prophylactic Vancomycin

SUMMARY:
This is a randomized 2-arm study to compare two different times of giving the drug vancomycin. Half of the patients will begin vancomycin two days before a bone marrow transplant. The other half will get it as soon as they have the first fever.

Streptococci are bacteria that live in one's mouth and gut. These bacteria can escape into the blood when the lining of the mouth and gut weakens from cancer therapy. This can make the person who is undergoing a bone marrow transplant very sick. All patients who get this infection are treated with antibiotics. Vancomycin is one drug that is used to treat this bloodstream infection once it is diagnosed. Studies have shown that giving vancomycin before a bone marrow transplant seems to prevent this infection. However, giving vancomycin too soon may increase the chance that the kidneys will be irritated. It may also increase the chance that other bacteria will become resistant to this drug. We, the investigators at Memorial Sloan-Kettering Cancer Center, do not know if waiting to start vancomycin until the patient has a first fever can also prevent this infection.

DETAILED DESCRIPTION:
The primary objective of this study is as follows:

* To compare prophylactic with empirical vancomycin administration for reducing early viridans streptococcal bacteremia in allogeneic hematopoietic stem cell transplant (HSCT) patients.

The secondary objectives of the study are:

* To examine the safety and tolerability for each vancomycin administration approach.
* To measure the incidence of vancomycin-resistant enterococcal (VRE) infections for patients managed with each of the two vancomycin administration approaches.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing allogeneic HSCT for hematologic malignancies or other disorders
* Conditioning regimen that includes high-dose total body irradiation (TBI) (>1200 cGy)
* The ability to understand and the willingness to sign the Institutional Review Board (IRB)-approved Informed Consent, including the Research Authorization component of the Informed Consent form.

Exclusion Criteria:

* Non-TBI conditioning regimen
* Prior history of hypersensitivity to vancomycin (excluding history of "Red Man Syndrome")
* Fever or infection that requires intravenous vancomycin or oral/intravenous linezolid between day-7 and day-3 before hematopoietic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126
Dates: Start 2003-11; Study Completion 2005-11

PRIMARY OUTCOMES:
To compare prophylactic with empirical vancomycin administration for reducing early viridans streptococcal bacteremia in allogeneic hematopoietic stem cell transplant (HSCT) patients

SECONDARY OUTCOMES:
To examine the safety and tolerability for each vancomycin administration approach
To measure the incidence of vancomycin-resistant enterococcal (VRE) infections for patients managed with each of the two vancomycin administration approaches

CONTACTS AND LOCATIONS:
Overall Officials: Susan Seo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org